CLINICAL TRIAL: NCT00176020
Title: Double-Blind, Randomized, Placebo-Controlled, Single-Center, 2 Treatment, 3-Way Crossover Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of a Single Oral Repeated Dose of 500 Mg Nicotinic Acid as Tablets in Healthy Subjects
Brief Title: Nicotinic Acid - Pharmacokinetics, Pharmacodynamics, Receptor Expression
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Other Study IDs: 2005-003234-18; K115
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-15 (Estimated); Status verified 2005-08

CONDITIONS: Healthy
Keywords: nicotinic acid; flush symptom; pharmacodynamic; pharmacokinetic
MeSH Terms: interventions — Niacin

INTERVENTIONS:
Drug: nicotinic acid

SUMMARY:
The study will be a double-blind, randomized, placebo-controlled, single-center, 2 treatment, 3--way crossover. Subjects will be randomly allocated to a treatment sequence - AAB, ABA or BAA. The two treatments will be:

* Treatment A: 500 mg nicotinic acid (Niacor(R))
* Treatment B: Niacor(R) Placebo

Each trial period will last one day, there will be a wash-out period of at least 2 days between each trial period. Five to seven days after study day 1 of trial period 3 there will be a final safety examination.

ELIGIBILITY:
Inclusion Criteria:

* Good state of health physically and mentally

Exclusion Criteria:

* Treatment with any other investigational product in the last 60 days before the day of randomization into the study
* Regular use of medication in the last 60 days before the day of randomization into the study except of oral contraceptives in female participants
* Treatment in the 60 days before the day of randomization into the study with any drug known to have a well-defined potential for toxicity to a major organ, or any substance which is known to induce or inhibit hepatic drug metabolism (including general anesthetics)
* Any drug intake (including over-the-counter remedies) in the 2 weeks before the day of randomization into the study, unless the investigator considers a drug intake to be clinically irrelevant for the purpose of this study
* Any acute or chronic illness or clinically relevant findings in the pre-study examination
* Presence, history or sequelae of gastrointestinal (e.g. peptic ulcer), liver or kidney disease, or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* History of hypersensitivity to the investigational product
* History or presence of abnormalities of the vascular bed
* History or presence of a dermatologic disease or skin lesions, particular in the area chosen for flush measurement
* History of allergy or hypersensitivity to other drugs or to food constituents
* History of other allergic diseases or hypersensitivity, unless the investigator considers it to be clinically irrelevant for the purpose of this study
* Blood donation of > 400 ml in the 60 days before the day of randomization into the study
* Smoking
* Positive result in urine screen for drugs of abuse or in alcohol breath test
* Known or suspected to be drug-dependent, including consumption of > 30 g alcohol per day
* Pregnancy or lactation
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, MD Bsc, Principal Investigator — Department Internal Medicine VI